CLINICAL TRIAL: NCT06894277
Title: Interactive Emotion Regulation Skills Training to Improve Adolescent Health Ph II
Brief Title: Internet-based Talking About Risk and Adolescent Choices: Health and Emotion Regulation Options
Acronym: iTRAC-HERO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Rhode Island Hospital (Other); University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0346; 4R42HD110333-02 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Risky Sexual Behavior; Emotion Regulation; Adolescent Behavior
Keywords: Risky Sexual Behavior; Emotion Regulation; Adolescent Behavior
MeSH Terms: conditions — Emotional Regulation; Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: Waitlist Control Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Waitlist Control (No Intervention): Control participants will be assessed on the same schedule as the treatment condition and offered the intervention after 6-month follow-up.
- iTRAC-HERO (Experimental): iTRAC-HERO is an 8-module, web-based intervention for middle school boys and girls to complete. Its goal is primary prevention of adolescent sexual risk behaviors by targeting emotion regulation and sexual self-efficacy. (e.g., to refuse sexual advances).
  Interventions: Behavioral: iTRAC-HERO

INTERVENTIONS:
Behavioral: iTRAC-HERO — iTRAC-HERO will consist of eight, approximately 45-minute, "gamified" digital modules of 4-6 activities (games, videos, etc.). No instruction is needed to use the program. Content will use gender- and sexuality-inclusive language and avoid heteronormative descriptions of risk. This content will include strategies for (and practice with) recognizing and managing emotions, particularly in relation to sexual health situations, to enhance the likelihood that the emotion regulation and sexual health education provided can be applied to experiences that are emotionally arousing and lead to risk.
  Arms: iTRAC-HERO

SUMMARY:
Using the efficacious iTRAC intervention to enhance emotion regulation competencies as a foundation, this study will create and test iTRAC-HERO to teach emotion regulation skills in the context of sexual health education.

DETAILED DESCRIPTION:
Adolescence is a critical developmental period during which behavioral patterns are formed that have powerful influences on current and future health. This is particularly true for sexual behavior, which is affected by the biological changes of puberty as well as normative developmental tasks around sexual exploration. Engaging in sexual behavior in early adolescence (before age 15) is associated with more partners, less condom use, and more frequent sex as teens get older, and these factors increase risk for negative health outcomes (e.g., sexually transmitted infections and unplanned pregnancy) throughout their lives. Many sexual health interventions teach prevention skills, such as assertiveness or condom use; the premise of the current application is that these skills are often unused by adolescents because of deficits in emotion regulation (ER), which is unaddressed in most sexual health education. Our research team has developed and tested a novel, engaging, efficacious, and developmentally tailored group intervention (Project TRAC) to teach ER skills to early adolescents within the context of sexual health. A study of Project TRAC showed that participants taught ER skills were less likely to start having sex over the 2.5 year follow up. While efficacious, the small group format of the Adolescence is a critical developmental period during which behavioral patterns are formed that have powerful influences on current and future health. This is particularly true for sexual behavior, which is affected by the biological changes of puberty as well as normative developmental tasks around sexual exploration. Engaging in sexual behavior in early adolescence (before age 15) is associated with more partners, less condom use, and more frequent sex as teens get older, and these factors increase risk for negative health outcomes (e.g., sexually transmitted infections and unplanned pregnancy) throughout their lives. Many sexual health interventions teach prevention skills, such as assertiveness or condom use; the premise of the current trial is that these skills are often unused by adolescents because of deficits in emotion regulation (ER), which is un-addressed in most sexual health education. The research team has developed and tested a novel, engaging, efficacious, and developmentally tailored group intervention (Project TRAC) to teach ER skills to early adolescents within the context of sexual health. A study of Project TRAC showed that participants taught ER skills were less likely to start having sex over the 2.5 year follow up. While efficacious, the small group format of the program presents barriers to sustainability and dissemination; significant advantages of web-based delivery exist. To explore whether the ER concepts of TRAC could be taught in a web-based format, the investigators completed a pilot study to translate TRAC's ER content to a web-based intervention (iTRAC), using Designing for Dissemination principles that enhance the likelihood of successful dissemination upon completion. iTRAC demonstrated feasibility and acceptability, and a randomized trial showed that iTRAC participants reported significantly better emotional competence compared to waitlist control participants. This study will complete the technology adaptation of the program to include its sexual health content and content linking ER to sexual health. This phase will create iTRAC-HERO as a web app. Once completed, acceptability testing will be completed with early adolescents to allow for modifications based on participant feedback. Once finalized, a small RCT will assess impact on adolescents' self-efficacy for preventing sexual risk as well as engagement in sexual behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Attending 7th grade
* Between 12 and 14 years old
* Parent/guardian speaks English or Spanish
* Attending participating school

Exclusion Criteria:

* Unable to read at a 4th grade level
* Have a sibling who has participated in the study
* Have a development disorder

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Change in Sexual Self-Efficacy (SSE) from baseline to 6 months. | Baseline, 1 month post-intervention, 6 month follow up
  The Sexual Self-Efficacy Scale (12 items) will measure self-efficacy for safer sexual activity as a main outcome which will indicate iTRAC-HERO's efficacy and ability to promote healthier sexual behaviors with the full sample (not just those who are sexually active).
Change in Self Efficacy for HIV Prevention from baseline to 6 month. | Baseline, 1 month post-intervention, 6 month follow up
  The Self-Efficacy for HIV Prevention Scale (12 items) assesses a range of behaviors related to prevention of HIV, other STIs, or unintended pregnancy, including refusing sexual behaviors, discussing sexual histories with partners, buying condoms, taking free condoms, carrying condoms, and asking a partner to use a condom.

SECONDARY OUTCOMES:
Change in Sexual Risk Cognition from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Sexuality Questionnaire for Adolescents (34 items) is a multiple choice test to assess sexual health knowledge and has been shown to be sensitive to intervention impact.
Change in attitudes towards abstinence from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Abstinence Attitudes questionnaire assesses agreement with values related to abstinence (α= .86).
Change in frequency of sexual and substance use behaviors from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Adolescent Risk Behavior Assessment (ARBA) will assess sexual behavior, including behaviors relevant to this developmental period.
Change in adolescent substance use behaviors from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  Youth Risk Behavior Surveillance System items will be used to assess tobacco/vape use, violence (e.g., fighting), and substance use behaviors.

OTHER OUTCOMES:
Change in Emotion Regulation Skills from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Difficulties in Emotion Regulation Scale (36 items) uses six subscales (e.g., lack of emotional awareness, limited access to ER strategies; all α > .80) to assess perceptions of skill in ER based on Linehan's theoretical work.
Change in frequency of dificulties with emotion regulation from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Affect Dysregulation Scale (6 items) assesses the frequency of difficulties with ER (α= .72), and is shown to be related to adolescent risk behaviors.
Change in usage of emotion regulation behaviors taught in iTRAC-HERO from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Emotion Regulation Behaviors Scale- Revised measures use of the specific emotion regulation strategies taught in iTRAC (α= .73).
Change in perceptions of one's ability to manage negative emotions from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Emotional Self-Efficacy Subscale of the Self-Efficacy Questionnaire for Children assesses perception of one's ability to cope with negative emotions (α= .83).
Change in beliefs about controllability of emotions from baseline to 6 months | Baseline, 1 month post-intervention, 6 month follow up
  The Implicit Theories of Emotions for Children Self subscale (6 items) is based on Dweck and colleagues' work on implicit theories of intelligence and Tamir's adult measure of emotion malleability. It assesses adolescents' beliefs about the controllability of their emotions (α=.86).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Houck, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Klein Buendel, Inc., Golden, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will prepare an archival-quality data package for upload to the National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH). Specifically, the investigators will provide documentation on the full data-audit trail from the exact prompts seen by participants, to the syntax used to score and aggregate items, to the finalized data ready for use by qualified investigators. The archival-quality data package will also include a codebook in line with the Data Documentation Initiative (DDI) and contains information about variables, metadata, and file structure. The metadata will include description of the trial, including design, implementation, and description of the interventions. The intent is to provide everything that future investigators require to understand the trial, analyze the data, correctly interpret the findings, and be able to publish new analyses that meet current publication standards for clinical trials and/or meta-analyses.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After analyses are completed for the aims of the study.
Access Criteria: The data package will be available for future investigators. For datasets that include potentially sensitive information, investigators not part of the original study will submit requests to be reviewed by the PIs. Qualified investigators who agree to terms of use and confidentiality agreements will be provided with deidentified data.